CLINICAL TRIAL: NCT07213362
Title: Study on the Effect of Different Doses of Computerized Cognitive Training on Cognitive Function in Patients With Mild Cognitive Impairment: An Open-Label, Randomized, Controlled Trial
Brief Title: Study on the Effect of Online Cognitive Training Doses on Cognitive Function in Individuals With Mild Cognitive Decline
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Haibo Wang, Research Fellow, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00001052-25101
Record Dates: First submitted 2025-09-16; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Disorder
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1: 30 min/session × 3 sessions/week (Active Comparator): CCT Training, 30 minutes per session, 3 times a week, for a total of 12 weeks
  Interventions: Device: Computerized Cognitive Training
- Group 2: 45 min/session × 5 sessions/week (Active Comparator): CCT Training, 45 minutes per session, 3 times a week, for a total of 12 weeks
  Interventions: Device: Computerized Cognitive Training
- Group 3: 60 min/session × 5 sessions/week (Active Comparator): CCT Training, 60 minutes per session, 3 times a week, for a total of 12 weeks
  Interventions: Device: Computerized Cognitive Training
- Group 4: 30 min/session × 5 sessions/week (Active Comparator): CCT Training, 30 minutes per session, 5 times a week, for a total of 12 weeks
  Interventions: Device: Computerized Cognitive Training
- Group 5: 45 min/session × 5 sessions/week (Active Comparator): CCT Training, 45 minutes per session, 5 times a week, for a total of 12 weeks
  Interventions: Device: Computerized Cognitive Training
- Group 6: 60 min/session × 5 sessions/week (Active Comparator): CCT Training, 60 minutes per session, 5 times a week, for a total of 12 weeks
  Interventions: Device: Computerized Cognitive Training

INTERVENTIONS:
Device: Computerized Cognitive Training — Computerized Cognitive Training (30 minutes per session, 3 sessions per week, for a 12-week period)
  Arms: Group 1: 30 min/session × 3 sessions/week
Device: Computerized Cognitive Training — Computerized Cognitive Training (45 minutes per session, 3 sessions per week, for a 12-week period)
  Arms: Group 2: 45 min/session × 5 sessions/week
Device: Computerized Cognitive Training — Computerized Cognitive Training (60 minutes per session, 3 sessions per week, for a 12-week period)
  Arms: Group 3: 60 min/session × 5 sessions/week
Device: Computerized Cognitive Training — Computerized Cognitive Training (30 minutes per session, 5 sessions per week, for a 12-week period)
  Arms: Group 4: 30 min/session × 5 sessions/week
Device: Computerized Cognitive Training — Computerized Cognitive Training (45 minutes per session, 5 sessions per week, for a 12-week period)
  Arms: Group 5: 45 min/session × 5 sessions/week
Device: Computerized Cognitive Training — Computerized Cognitive Training (60 minutes per session, 5 sessions per week, for a 12-week period)
  Arms: Group 6: 60 min/session × 5 sessions/week

SUMMARY:
The primary questions that this clinical trial aims to answer are:

To compare the differences in the efficacy of different doses of Computerized Cognitive Training (CCT) in improving cognitive function among patients with Mild Cognitive Impairment (MCI), and to explore the potential optimal intervention dose.

To analyze the interaction between individual characteristics and the intervention dose of CCT.

To compare the improvement in functional activity ability of MCI patients among different CCT intervention dose groups.

To compare the symptoms of depression and anxiety among different CCT intervention dose groups.

To evaluate the adherence to different doses of CCT intervention.

Participants will:

Receive CCT intervention at varying durations and frequencies over a 12-week period, and will be followed up for cognitive function, functional activity ability, etc., at weeks 4, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years.
* Self-reported cognitive decline, confirmed by an informant.
* Montreal Cognitive Assessment (MoCA) score of 19-25, adjusted for years of education (+1 point for 12 years or less).
* Ability to complete activities of daily living independently.
* Possesses basic communication skills and is able to cooperate with the study procedures.
* Voluntarily agrees to participate in the study and signs the informed consent form.

Exclusion Criteria:

* Presence of underlying neurological diseases that may impair cognitive function, including but not limited to dementia syndrome, Parkinson's disease, epilepsy, and cerebrovascular disease.
* Presence of severe or unstable organic diseases such as cancer, hydrocephalus, history of central nervous system tumors, or acute brain injury/infection.
* Diagnosis of severe mental illness such as major depressive disorder, schizophrenia, schizoaffective disorder, or bipolar disorder.
* Presence of severe visual or hearing impairment, or other physical conditions that may interfere with the completion of the study.
* Participation in any other clinical trial within the past 3 months.
* Having received transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), light therapy, or having taken medications that could significantly affect cognitive function (e.g., nootropics, psychoactive drugs, anticholinergic drugs, benzodiazepines) for any reason within the past 6 months.
* History of alcohol dependence or substance abuse.
* Consumption of alcohol or other substances that affect cognitive function, such as caffeine or cocaine, within 24 hours prior to the cognitive assessment.

Any other conditions that the investigator deems unsuitable for participation in this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The improvement in cognitive function from baseline at week 12 post-randomization, assessed by the Montreal Cognitive Assessment (MoCA) total score. | Week 12 post-randomization
  Scores derived from this assessment scale range from 0 to 30. A higher score corresponds to superior cognitive ability.

SECONDARY OUTCOMES:
Mental health status at weeks 4, 12, and 24 post-randomization, assessed using the Patient Health Questionnaire-4 (PHQ-4) | Weeks 4, 12, and 24 post-randomization.
  Scores derived from this assessment scale range from 0 to 12. A higher score corresponds to worse mental health status.
Cognitive performance in sub-domains at weeks 4, 12, and 24 post-randomization, assessed based on the cognitive index, which is calculated by the cognitive training platform using scores from the training process. | Weeks 4, 12, and 24 post-randomization.
Functional activities at weeks 4, 12, and 24 post-randomization，assessed based on the scores from the Functional Activity Questionnaire(FAQ) | at weeks 4, 12, and 24 post-randomization.
  Scores derived from this assessment scale range from 0 to 30. A higher score corresponds to superior functional activity ability.
Change from baseline in Montreal Cognitive Assessment (MoCA) scale scores at weeks 4 and 24 post-randomization. | Weeks 4 and 24 post-randomization
  Scores derived from this assessment scale range from 0 to 30. A higher score corresponds to superior cognitive ability.

OTHER OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | at weeks 4, 12, and 24 post-randomization.

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code